CLINICAL TRIAL: NCT01805687
Title: A Single-Center, Open-Label, Single-Dose Evaluation of the Duration and Extent of Bronchodilation Following Administration of Zileuton CR 1200 mg in Subjects With Stable, Chronic Asthma
Brief Title: Single Dose Bronchodilatory Study in Asthma
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cornerstone Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRTX 082-04-01
Record Dates: First submitted 2013-03-05; First posted 2013-03-06 (Estimated); Results first posted 2014-08-18 (Estimated); Last update posted 2014-09-03 (Estimated); Status verified 2014-08

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

ARMS (1):
- Zileuton extended release (Other): Oral, 1200 mg (2 x 600 mg tablets)
  Interventions: Drug: Zileuton extended release

INTERVENTIONS:
Drug: Zileuton extended release

SUMMARY:
Study to evaluate the bronchodilator effects of Zyflo CR in patients with chronic stable asthma.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of asthma for at least 5 years
* FEV1 of 50-85% predicted
* Reversible airway obstruction

Exclusion Criteria:

* Pregnant/nursing females
* Liver function tests greater than upper limit of normal

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2013-03; Primary Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Northeast Medical Research Associates, North Dartmouth, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Zileuton Extended Release: Zileuton extended release 1200 mg (2 x 600 mg tablets)
Period: Overall Study
Arm/Group | Zileuton Extended Release
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Zileuton Extended Release: Zileuton extended release
Arm/Group | Zileuton Extended Release
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 35 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 8

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in FEV1
Time Frame: 12 Hours
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | Zileuton Extended Release
Number analyzed (Participants) | 25
Liter | 2.84 (0.706)

2. Secondary Outcome: Area Under the Curve (AUC)
Time Frame: 72 Hours
Reporting Status: Not Posted

3. Secondary Outcome: Number of Subjects With Adverse Events
Time Frame: 72 Hours
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Zileuton Extended Release
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 3/25
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zileuton Extended Release (N=25)
Abnormal Liver Function (Hepatobiliary disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less